CLINICAL TRIAL: NCT01410643
Title: Puberty Related Intervention to Improve Metabolic Outcomes (The PRIMO Study)
Acronym: PRIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UAB
Record Dates: First submitted 2011-03-30; First posted 2011-08-05 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: puberty; body composition; metabolism; obesity; optimization of body composition; pubertal transition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced Carbohydrate (Active Comparator): 42% carbohydrate macronutrient modification
  Interventions: Other: Macronutrient Modification
- STandard Carbohydrate (Active Comparator): 60% carbohydrate macronutrient modification
  Interventions: Other: Macronutrient Modification

INTERVENTIONS:
Other: Macronutrient Modification — reduced carbohydrate versus standard carbohydrate diet

SUMMARY:
Puberty represents a critical period in terms of metabolic health. Racial differences in insulin dynamics, reproductive maturation, and the associated endocrine changes may affect a female's health later in life. Further, the peripubertal period is likely the period of racial divergence in adiposity noted between European American (EA) and African American (AA) girls. Diet is a major modifiable risk factor. The identification of simple, cost-effective dietary strategies for prevention and management of metabolic disease and excess fat mass accrual during the peripubertal period is a priority. Modification of the diet to affect metabolic and endocrine outcomes with and without weight loss during the pubertal transition represents a novel approach to the pediatric obesity epidemic.

It is likely that the two diets used in this project will have different metabolic effects, including effects on postprandial glycemia, triglyceride concentration, free fatty acid concentration, and satiety. These factors may in turn, affect development of metabolic perturbations, especially in susceptible individuals (e.g. AA peripubertal girls).The role of carbohydrates on metabolic outcomes, particularly among children, has received little attention. It has been hypothesized that higher postprandial glycemia may be a mechanism for disease progression. Development of a diet that reduces insulin secretion and optimizes metabolic-endocrine health among peripubertal girls will likely reduce obesity and related co-morbidities and future reliance on pharmacologic treatments, even in the absence of weight loss. However, in light of the current trends in pediatric obesity, a safe and effective regimen that also promotes weight loss is needed for the pediatric population.

This proposal is significant in that it will shed light on whether diet composition, as a part of a eucaloric (weight-stable) or hypocaloric diet (weight-loss) can influence the hyperinsulinemic characteristic of AA peripubertal girls. Existing data suggest that elevated concentrations of insulin and/or reproductive hormones may contribute to the fat mass accrual in AA and could elevate risks for development of chronic diseases in adulthood. The results of this study will lead to the development of dietary means for the reduction of insulin, and thereby to the prevention of both pediatric obesity and type 2 diabetes.

DETAILED DESCRIPTION:
This study will include 100 European and African American girls ages 7-11 years. Subjects must be non-diabetic and overweight (percentile BMI >85th ).

Screening First they will complete a telephone questionnaire regarding medical history and current lifestyle (approximately 15 minutes). If the subject is deemed eligible based on the telephone screening, they will come to UAB for an orientation meeting. At this time the subjects' height and weight will be recorded. They will receive a copy of the study assent/consent form and review the entire protocol with selected study personnel (approximately 60 minutes).

Protocol

Run-In Phase With parental guidance, subjects will complete a 4-day food record for assessment of typical nutrient intake (attached) prior to beginning the run-in diet. The 4-day food record will be analyzed by a registered dietitian using the Minnesota Nutrition Data System. Then subjects will be provided food for 3 days. This diet is similar to the standard "American" diet, and is intended to eliminate inter-subject variance in metabolic outcomes due to free-living dietary factors. The total energy of all diets will be calculated to be eucaloric so that body weight is maintained, and will be determined using the Harris-Benedict equation with an activity factor of 1.35. In previous and ongoing studies at the UAB CRU, this method has resulted in maintenance of body mass. Subjects will come to UAB to be weighed and pick up meals. All meals will be packaged for home consumption. Upon completion of the Run-in Phase, subjects will report to the CRU Outpatient facilities for metabolic testing and WEBB and Boshell buildings for body composition assessment. The tests administered are described below.

Phase 1 Weeks 1-6. Subjects will be randomized to a controlled eucaloric reduced-CHO (SPEC) or a controlled eucaloric standard (STAN) diet. Subjects will come to UAB two days a week in the morning (Monday-Friday) to be weighed and to collect food for their meals. Energy needs will be estimated by a qualified dietitian using standard equations. All foods for the diet intervention will be provided by the study. Body weight will be recorded to ensure weight maintenance. Energy intake will be adjusted if necessary to maintain body weight. Upon completion, subjects will report to the CRU Outpatient facilities for metabolic testing and WEBB building for body composition assessment. The tests administered are described in the chart below.

One morning, approximately at the midpoint of phase 1, subjects will be asked to come to the CRU and undergo a solid meal test. This test will measure the hormonal and glycemic response to consuming a breakfast that will be provided as a part of the study. The details of this test are outlined below.

Phase 2 Weeks 7-18. Subjects will continue in their assigned diet groups (i.e. SPEC or STAN), but will now receive a controlled hypocaloric diet designed to facilitate weight loss. Subjects will report to UAB two weekday mornings to be weighed and to collect food for their meals. Energy needs will be estimated by a qualified dietitian. All foods for the diet intervention will be provided by the study. Body weight will be recorded two times weekly to monitor weight loss. Upon completion of phase 2, subjects will report to the CRU Outpatient facilities for metabolic testing and the WEBB building for body composition assessment. The tests administered are described in the chart below.

Education and Counseling Sessions At the time of completion of Phase 2, study participants will initiate a series of education and counseling sessions designed to allow them to continue with their assigned diets under a free-living situation for the ensuing 6 weeks. The goal of this phase will be maintenance of the weight loss that occurred during the formal intervention. Subjects will attend group meetings during the 6-week follow-up phase. These meetings will occur weekly during weeks 19-22, and bi-weekly during weeks 23-25. The periodic education and counseling sessions will serve to reinforce the diet guidelines, and to evaluate any problems that have arisen.

Phase 3 Weeks 19-25 subjects will be in a "free-living phase." During weeks 19-25, a dietitian will periodically administer unannounced 24-hour diet recalls by telephone. This involves subjects reporting foods they consumed during the previous day. At the end of Phase 3 subjects will receive a DXA scan and have resting energy expenditure assessed.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as African American or European American
* Aged 7-11 AND Tanner stage < 3
* Overweight (BMI percentile 85-97th)
* Not taking any medication known to affect body composition
* No prior diagnosis of chronic condition

Exclusion Criteria:

* Illness that precludes study participation
* Prescribed medication known to affect body composition
* Not of EA or AA racial/ethnic group
* Obese (BMI% > 97th) or normal weight (BMI% < 85th)
* Reproductively mature as define by Tanner stage > 3

Ages: 7 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Determine if a hypocaloric (weight-loss), SPEC diet results in greater fat loss than a 12-week, hypocaloric, STAN diet among overweight females aged 7-11 years. | 12-weeks
  The SPEC diet will be more effective than the STAN diet at promoting fat loss (while preserving bone mass). Evaluate insulin sensitivity, insulin secretion, reproductive hormone status, resting energy expenditure compared to baseline.
  Outcomes will be assessed in serum by measurement of insulin/glucose following a liquid meal tolerance test and whole-body body composition bone marrow adipose tissue volume (cm^3); trabecular bone (g) via DXA, MRI, and pQCT, respectively. We will evaluate changes in estradiol (pg/ml), FSH (pg/ml), LH (pg/ml), testosterone (pg/ml) and lipid profile.

SECONDARY OUTCOMES:
To evaluate the relationship between genetic factors and the physiologic, hormonal, and metabolic response to the two diets, the genetic admixture and genetic association will be evaluated. | 16 weeks
  The SPEC diet will be more effective than the STAN diet in decreasing insulin secretion and increasing insulin sensitivity. The SPEC diet will be more effective in reducing insulin, which in turn will reduce estradiol (or the estrogen-androgen ratio) and thereby minimize the relative gain in fat mass.
  Evaluate changes in insulin sensitivity, insulin secretion, reproductive hormone concentration, resting energy expenditure and body composition from baseline and compare results between two arms.
Determine if a low-carbohydrate diet (SPEC) is more effective than a standard (STAN) diet in decreasing insulin secretion, increasing insulin sensitivity, and decreasing estradiol concentration among overweight girls 7-11 years. | 6-weeks
  This outcome aims to evaluate metabolic and endocrine changes that occur in the absence of weight change.

CONTACTS AND LOCATIONS:
Overall Officials: Krista R Casazza, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Hanks LJ, Gutierrez OM, Ashraf AP, Casazza K. Bone Mineral Content as a Driver of Energy Expenditure in Prepubertal and Early Pubertal Boys. J Pediatr. 2015 Jun;166(6):1397-403. doi: 10.1016/j.jpeds.2015.02.054. Epub 2015 Apr 1. PMID 25841541